CLINICAL TRIAL: NCT07359651
Title: Factors Associated With In-hospital Mortality in Necrotizing Soft Tissue Infections. A Multicenter Retrospective Cohort Study. FATAL-NSTI Study (Factors Associated With In-hospital mortALity in NSTI).
Brief Title: FATAL-NSTI Study (Factors Associated With In-hospital mortALity in NSTI).
Acronym: FATAL-NSTI
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: University of Cagliari, Cagliari, Italy (Unknown); University of Milano Bicocca (Other); University of Milan (Other); Università Cattolica del Sacro Cuore, Rome, Italy (Unknown)
Responsible Party: Principal Investigator, Mauro Podda, Professor, University of Cagliari
Other Study IDs: FATAL-NSTI_UniCa_2025.
Record Dates: First submitted 2026-01-07; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Necrotizing Fascitis; Fournier Gangrene; Fournier's Gangrene; Soft Tissue Infections
Keywords: Necrotizing soft tissues infections; NSTI; Necrotizing fasciitis; Fournier's gangrene
MeSH Terms: conditions — Fasciitis, Necrotizing; Fournier Gangrene; Soft Tissue Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with Necrotizing Soft Tissue Infections.: Adult patients admitted with a diagnosis of necrotizing soft tissue infection, diagnosed based on clinical findings, imaging when available, and/or intraoperative assessment.
  Interventions: Other: No Intervention: Observational Cohort
- Necrotizing Fasciitis: Patients with necrotizing infection primarily involving the fascia and surrounding soft tissues, diagnosed based on clinical findings, imaging when available, and/or intraoperative assessment.
  Interventions: Other: No Intervention: Observational Cohort
- Fournier's Gangrene: Patients with necrotizing infection involving the perineal, genital, or perianal region, consistent with Fournier's gangrene.
  Interventions: Other: No Intervention: Observational Cohort
- Necrotizing Soft Tissue Infections of the Neck and Trunk: Patients with necrotizing soft tissue infections involving the cervical region or the trunk, including thoracic and abdominal wall locations.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No experimental intervention, treatment assignment, or change in clinical management is performed as part of the study.
  All patients receive standard medical and surgical care according to local institutional protocols and current clinical practice guidelines. Diagnostic and therapeutic decisions are made solely by the treating clinical teams and are not influenced by participation in the study.

SUMMARY:
Necrotizing soft tissue infections (NSTIs) are rare but potentially life-threatening infections involving the skin and underlying tissues such as fat, fascia, and sometimes muscle. They can progress rapidly and, despite modern antibiotics, surgery, and intensive care, are still associated with high in-hospital mortality.

A major challenge in the management of NSTIs is early diagnosis. Initial signs and symptoms are often nonspecific and may resemble less severe soft tissue infections, leading to diagnostic and therapeutic delays. Once identified, treatment requires urgent surgery, broad-spectrum antibiotics, and close monitoring, frequently in an intensive care setting.

Even with appropriate treatment, the clinical course of NSTIs is highly variable. Some patients recover, while others develop severe complications such as septic shock or multiple organ failure and may die during hospitalization. Predicting outcomes early in the hospital stay remains difficult for clinicians.

The aim of this observational study is to identify factors associated with in-hospital mortality in adult patients with NSTIs. In-hospital mortality, defined as death from any cause during the hospital stay for NSTI treatment, represents the most severe outcome and is of major relevance to patients and caregivers.

The study focuses on clinical and laboratory data routinely available at hospital admission or during initial emergency department evaluation. These include patient demographics, vital signs, and standard blood test results commonly obtained in early clinical assessment. No additional diagnostic tests or procedures are required for study purposes.

Identifying early predictors of mortality is particularly important in NSTIs, given the rapid progression of the disease. Early recognition of high-risk patients may allow closer monitoring and more timely interventions.

The study will be conducted in high-volume referral centers with extensive experience in NSTIs management, where care is delivered according to established international guidelines. All patients will receive standard treatment based on clinical judgment. No experimental therapies or changes in routine care will be involved.

DETAILED DESCRIPTION:
Necrotizing soft tissue infections (NSTIs) represent a group of rare but extremely severe conditions characterized by rapid progression, extensive tissue destruction, and a high risk of systemic complications. These infections often require surgical management in emergency settings, broad-spectrum antimicrobial therapy, and intensive supportive care. Despite improvements in diagnostic strategies, surgical techniques, and critical care, NSTIs continue to be associated with high in-hospital mortality and substantial morbidity.

The main clinical challenge in the management of these infections is the difficulty in predicting outcomes early in the hospital course. Initial signs and symptoms may be nonspecific and can overlap with those of less severe soft tissue infections. Early risk assessment remains complex, particularly during the first hours after hospital admission, when critical decisions regarding monitoring intensity, resource allocation, and escalation of care must be made.

The present study is designed to improve understanding of factors associated with adverse outcomes in patients with NSTIs by focusing on clinical and laboratory information available at the time of hospital admission. The study aims to identify early indicators of increased risk that can be recognized promptly in everyday clinical practice through the analysis of variables routinely collected during initial evaluation.

The study involves four tertiary referral academic hospitals in Italy, all of which are high-volume centers with extensive experience in the management of NSTIs and other (traumatic and septic) complex surgical emergencies.

Data used for this study are derived from routinely collected clinical information recorded during standard patient care. The dataset includes demographic characteristics, comorbid conditions, physiological parameters, and laboratory test results obtained at hospital admission and during the initial clinical assessment. The selected variables are widely available, rapidly obtainable, and commonly used by clinicians to evaluate patient status at presentation.

The study aims to clarify how combinations of early clinical and laboratory findings are associated with death and other severe in-hospital outcomes.

The study does not seek to influence or modify clinical management but rather to provide prognostic information that may complement clinical judgment.

The analytical approach includes exploratory and confirmatory statistical analyses to assess associations between admission variables and adverse outcomes. Multivariable modeling techniques are used to account for the combined effect of multiple factors and to identify independent predictors of poor outcomes.

The results of the multivariable model will be translated into a graphical risk estimation tool. This tool is intended to provide an intuitive representation of how different admission variables contribute to overall risk.

All data are handled in accordance with applicable ethical standards and data protection regulations. The study uses retrospective data collected during routine care, and appropriate approvals were obtained from institutional authorities at each participating center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Hospital admission with a diagnosis of necrotizing soft tissue infection, including: Necrotizing fasciitis, Fournier's gangrene, Necrotizing soft tissue infections involving the neck or trunk.

Exclusion Criteria:

* Age younger than 18 years
* Patients with non-necrotizing skin or soft tissue infections
* Patients transferred to another hospital before completion of treatment or outcome assessment
* Missing data for the primary outcome (in-hospital mortality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients admitted to the participating high-volume tertiary referral academic hospitals in Italy with a diagnosis of necrotizing soft tissue infection. Patients are managed according to standard clinical practice by experienced multidisciplinary teams, including emergency surgeons, trauma surgeons, and critical care specialists. The population includes patients affected by different forms of necrotizing soft tissue infections, such as necrotizing fasciitis, Fournier's gangrene, and necrotizing infections involving the neck or trunk. All patients are evaluated and treated during the index hospitalization, and clinical data are collected as part of routine medical care. Only information available at the time of hospital admission or during the initial clinical assessment is used for analysis.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days from hospital admission.
  Death from any cause occurring during the index hospitalization for necrotizing soft tissue infection.

SECONDARY OUTCOMES:
Limb amputation (upper or lower extremity) | 30 days from hospital admission.
  Need for surgical amputation of the upper or lower limb performed during the index hospitalization for necrotizing soft tissue infection.

CONTACTS AND LOCATIONS:
Overall Officials: Adolfo Pisanu, MD, Study Director — University of Cagliari
Locations (4):
- Italy (4):
  - Cagliari University Hospital "Duilio Casula"., Cagliari
  - Niguarda Hospital, Trauma team., Milan
  - San Gerardo Hospital, Department of Surgery, Monza
  - Gemelli Hospital, Rome. Department of Surgery., Roma

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Data sharing is restricted due to patient confidentiality, data protection regulations, and local institutional policies.